CLINICAL TRIAL: NCT03957785
Title: Lower Body Positive Pressure Treadmill Training in Post-Stroke Gait Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Rocco Salvatore Calabrò, Clinical Professor, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRCCSME 19/2017
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Gait, Hemiplegic
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alter G treatment (Experimental): All participants practiced one session a day of AlterG (for 40min), six days a week, for four weeks (for a total amount of 24 sessions). All patients were trained using BWS, and treadmill speed (S) to allow the participant to walk with the intermittent support of one physiotherapist to help with balance and coordination. A qualitative (using FAC) and quantitative (spatio-temporal parameters and dynamic electromyography) gait assessment before and after the end of the gait training was performed.
  Interventions: Device: AlterG Treatment
- Traditional Gait Training (Active Comparator): All participants practiced one session a day TGT (for 40min), six days a week, for four weeks (for a total amount of 24 sessions). All patients were trained using FAC-tailored physiotherapist assistance, to allow the participant to walk with the intermittent support of one physiotherapist to help with balance and coordination (FAC 2), with the visual supervision of one physiotherapist (FAC 3), or independently without using the handrails (FAC 4). Physiotherapist assistance, and S were checked and adapted to subjects' progresses across the AlterG sessions.
  Interventions: Device: AlterG Treatment
- Healthy Control (Active Comparator): ll participants practiced one session a day of AlterG (for 40min), six days a week, for four weeks (for a total amount of 24 sessions). All patients were trained using BWS, and treadmill speed (S) to allow the participant to walk with the intermittent support of one physiotherapist to help with balance and coordination. A qualitative (using FAC) and quantitative (spatio-temporal parameters and dynamic electromyography) gait assessment before and after the end of the gait training was performed.The HC initially practiced the device at the same BWS and S administered to the patients. BWS and S were reduced progressively and increased, respectively, across the AlterG sessions in keeping with patients progresses.
  Interventions: Device: AlterG Treatment

INTERVENTIONS:
Device: AlterG Treatment — All participants practiced one session a day of AlterG or TGT (for 40min), six days a week, for four weeks (for a total amount of 24 sessions). All patients were trained using BWS, FAC-tailored physiotherapist assistance, and treadmill speed (S) to allow the participant to walk with the intermittent support of one physiotherapist to help with balance and coordination (FAC 2), with the visual supervision of one physiotherapist (FAC 3), or independently without using the handrails (FAC 4). BWS, physiotherapist assistance, and S were checked and adapted to subjects' progresses across the AlterG sessions. A qualitative (using FAC) and quantitative (spatio-temporal parameters and dynamic electromyography) gait assessment before and after the end of the monthly LBPP gait training was carried out.

SUMMARY:
Lower body positive pressure (LBPP) decreases weight bearing and ground reaction forces, with potentially positive effects on qualitative gait indices. However, which gait features are shaped by LBPP gait training in post-stroke patients is still poorly predictable. A pilot study on the effects of LBPP gait training on qualitative and quantitative gait indices in patients with hemiparesis due to stroke in the chronic phase was carried out. Twenty-five patients who suffered from a first, single, ischemic, supra-tentorial stroke occurred at least 6 months before study inclusion were provided with 24 daily sessions of LBPP treadmill gait training using AlterG device. These patients were compared with 25 age-matched healthy controls (HC), who were formerly provided with the same amount of AlterG training, and 25 patients with the same clinical-demographic characteristics of the first group of patients, who previously underwent conventional treadmill gait training (TGT). Qualitative and quantitative gait features, including Functional Ambulation Categories, gait cycle features, and muscle activation patterns were analyzed before and after the training (AlterG or TGT).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 55 years;
* first, single, ischemic supra-tentorial stroke occurred at least 6 months before the study inclusion;
* a Functional Ambulatory Categories (FAC) score of >2;
* ability to control head and trunk posture;
* no systemic or cardiovascular contraindication to LBPP

Exclusion Criteria:

• Medical and/or psychiatric illness potentially interfering with the treatment.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Functional Ambulatory Categories | 1 month
  FAC is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device

SECONDARY OUTCOMES:
gait cycle duration | 1 month
  GCD is the time interval between two successive occurrences of one of the repetitive events of walking, herein the right heel strike),

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided